CLINICAL TRIAL: NCT02290392
Title: The Minority Health Genomics and Translational Research BIo-Repository Database (MH-GRID)-2.0
Brief Title: Minority Health Genomics and Translational Research Bio-Repository Database (MH-GRID)-2.0
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999915011; 15-HG-N011
Record Dates: First submitted 2014-11-11; First posted 2014-11-14 (Estimated); Last update posted 2025-12-08 (Actual); Status verified 2025-10-01

CONDITIONS: Hypertension
Keywords: African American; Natural History
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: African Americans age 30-55 years with severe controlled HTN or severe resistant HTN.

SUMMARY:
Background:

- High blood pressure is a common problem. It can cause heart attacks, strokes, and kidney failure. It affects African Americans more than other racial groups. Data were collected from over a thousand African Americans across the country. The data were put into a database (MH-GRID). The data were about genes, diet, sleep, body mass index. They also cover stress and access to healthy foods and parks. Researchers at NIH will study these data in new ways. They want to learn more about the connection between African Americans and high blood pressure.

Objective:

- To study MH-GRID data to find the causes of severe high blood pressure and other cardio-metabolic problems in people of African ancestry.

Eligibility:

- African Americans age 30 55 with severe high blood pressure were used in the MH-GRID study. No new participants will be enrolled in this study.

Design:

- Researchers will examine data from the MH-GRID study.

DETAILED DESCRIPTION:
The etiology of racial/ethnic differences in health involves dynamic interactions between

genetic, behavioral and social-environmental determinants. Despite this, the field lacks robust

datasets that integrate these determinants with clinical assessments in minority patient cohorts. The Minority Health Genomics and Translational Research Bio-repository Database (MHGRID) Network infrastructure facilitated the collection of biospecimens and related multidimensional data elements within a consortium of minority-serving clinics. This initiative expands the diversity of ancestral groups in national genomic medicine datasets and promises to accelerate the translation of personalized medicine into minority communities. The MH-GRID project was initiated by Dr. Gibbons (founding PI) prior to becoming an NIH investigator. The MH-GRID project has completed its participant recruitment activities, closed out its NIH funding and now represents an existing dataset and biorepository that is being transferred to NHLBI for ongoing secondary analyses. A variety of investigations will be conducted on this existing dataset. The primary outcome variables include severe hypertension and hypertension induced kidney damage. Secondary outcome variables include obesity, coronary heart disease and metabolic disease syndrome. Intervening variables include genetics, behavioral (i.e. sleep quality, health literacy, smoking, diet, body mass index), ancestry, social (i.e. socioeconomic status, racial discrimination, stress, social deprivation), biological (i.e. insulin resistance, cholesterol, inflammatory markers), and environmental (i.e. neighborhood, access to healthy foods, parks).

ELIGIBILITY:
* INCLUSION CRITERIA:
* The MH-GRID Project s inclusion criteria included AA age 30-55 years
* Severe controlled HTN or severe resistant HTN

EXCLUSION CRITERIA:

* Exclusion criteria involved patients with secondary forms of HTN, primary forms of kidney disease or major co-morbidities (e.g. diabetes, heart failure, end-stage renal failure, HIV, and liver disease)
* Children <18 were not enrolled in the protocol

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Sampling Method: Non-Probability Sample
Enrollment: 1692 (Actual)
Dates: Start 2014-11-11; Primary Completion 2019-07-16 (Actual); Study Completion 2019-07-16 (Actual)

PRIMARY OUTCOMES:
To complete the original MH-GRID primary outcome analyses by defining the genetic, behavioral , and social-environmental determinants of severe hypertension and other cardio-metabolic disorders in individuals of African ancestry. | one time analysis
  To complete the original MH-GRID primary outcome analyses by defining the genetic, behavioral , and social-environmental determinants of severe hypertension and other cardio-metabolic disorders in individuals of African ancestry.

SECONDARY OUTCOMES:
The secondary outcome variables include obesity, coronary heart disease and metabolic disease syndrome. Intervening variables include genetics, behavioral, ancestry, social, biological, and environmental. | one time analysis
  The secondary outcome variables include obesity, coronary heart disease and metabolic disease syndrome. Intervening variables include genetics, behavioral, ancestry, social, biological, and environmental.

CONTACTS AND LOCATIONS:
Overall Officials: Tiffany M Powell-Wiley, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Heart, Lung and Blood Institute (NHLBI), Bethesda, Maryland, United States